CLINICAL TRIAL: NCT03919032
Title: Bacterial Infections in Patients with Cirrhosis in Argentina
Brief Title: Bacterial Infections in Patients with Cirrhosis in Argentina: Clinical and Microbiological Characteristics
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, SEBASTIAN MARCIANO, Assistant Professor of Hepatology , Principal Investigator, Hospital Italiano de Buenos Aires
Other Study IDs: 3879
Record Dates: First submitted 2019-04-10; First posted 2019-04-18 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2020-02

CONDITIONS: Bacterial Infections; Cirrhosis; Resistant Infection; Morality
MeSH Terms: conditions — Bacterial Infections; Fibrosis | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: This is an observational study without intervention — This is an observational study without intervention

SUMMARY:
In recent years, there has been an increasing prevalence of bacterial infections caused by multiresistant and extremely resistant organisms in patients with cirrhosis. These infections are associated with a worse prognosis, generate difficulties in the management of the patient during hospitalization and increase health costs.

The main objective of this project is to estimate the prevalence of infections by multiresistant bacteria in patients with cirrhosis. Additionally, the prevalence of other antibiotic resistance patterns and morbi-mortality in the study population will be evaluated.

For these purposes, a multicenter prospective cohort study will be carried out, including patients with cirrhosis who present bacterial infections at the time of admission, or during hospitalization.

Performing a study in Argentina on the clinical and microbiological characteristics of bacterial infections in patients with cirrhosis could be very useful to develop new strategies for prevention and treatment of this severe complication.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis
* Patients older than 17 years.
* Patients who are hospitalized for bacterial infections, or who develop bacterial infections while hospitalized

Exclusion Criteria:

• Refusal to participate in the informed consent process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 17 years with cirrhosis who are hospitalized for bacterial infections, or who develop bacterial infections while hospitalized
Sampling Method: Probability Sample
Enrollment: 472 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
To estimate the prevalence of infections caused by multi-resistant microorganisms in patients with cirrhosis | at the moment of the diagnosis of the bacerial infection

SECONDARY OUTCOMES:
To evaluate variables associated with infections caused by multi-resistant microorganisms in patients with cirrhosis | at the moment of the diagnosis of the bacerial infection
To evaluate the effect of infections caused by multi-resistant microorganisms on the in-hospital survival of patients with cirrhosis | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Sebastián Marciano, Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vazquez C, Gutierrez-Acevedo MN, Barbero S, Notari LDC, Agozino M, Fernandez JL, Anders MM, Grigera NL, Antinucci F, Orozco-Ganem ONF, Murga MD, Perez MD, Palazzo AG, Rejtman LM, Duarte IG, Vorobioff JD, Trevizan V, Bulaty S, Bessone F, Valverde M, Elizondo M, Borzi SM, Stieben TE, Masola AC, Ferretti SE, Arufe D, Demirdjian E, Raffa MP, Peralta M, Fainboim HA, Vazquez CE, Ruiz PM, Martinez JE, Heffner LA, Odzak A, Dirchwolf M, Smud A, Mendizabal M, Calzetta PA, Martinez A, Tomatis J, Bruno A, Ramos A, Pages J, Tevez S, Gadano AC, Giunta DH, Marciano S. Clinical and microbiological characteristics of bacterial infections in patients with cirrhosis. A prospective cohort study from Argentina and Uruguay. Ann Hepatol. 2023 Jul-Aug;28(4):101097. doi: 10.1016/j.aohep.2023.101097. Epub 2023 Apr 6. PMID 37030570
- [Derived] Marciano S, Gutierrez-Acevedo MN, Barbero S, Del C Notari L, Agozino M, Fernandez JL, Anders MM, Grigera N, Antinucci F, Orozco Ganem OF, Murga MD, Perez D, Palazzo A, Martinez Rejtman L, Duarte IG, Vorobioff J, Trevizan V, Bulaty S, Bessone F, Valverde M, Elizondo M, Bosia JD, Borzi SM, Stieben TE, Masola A, Ferretti SE, Arufe D, Demirdjian E, Raffa MP, Peralta M, Fainboim HA, Vazquez CE, Ruiz P, Martinez JE, Heffner LA, Odzak A, Dirchwolf M, Smud A, Mendizabal M, Bellizzi C, Martinez A, Tomatis J, Bruno A, Ramos A, Pages J, Tevez S, Gadano AC, Giunta DH. Norfloxacin prophylaxis effect on multidrug resistance in patients with cirrhosis and bacterial infections. Eur J Clin Microbiol Infect Dis. 2023 Apr;42(4):481-491. doi: 10.1007/s10096-023-04572-2. Epub 2023 Feb 23. PMID 36820931